CLINICAL TRIAL: NCT04228055
Title: Comprehensive Lifestyle Improvement Program for Men With Prostate Cancer2 (CLIPP2)
Acronym: CLIPP2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1806697620-2
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: Low Carbohydrate; Ketogenic; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Pre and Post Study Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLIPP2 (Experimental): 24 Week Lifestyle Modification Intervention
  Interventions: Behavioral: CLIPP2

INTERVENTIONS:
Behavioral: CLIPP2 — Diabetes Prevention Program and Comprehensive Lifestyle Improvement Program with emphasis on a low carbohydrate and Keto diet, physical activity, sleep optimization and stress management.

SUMMARY:
This study is an investigator initiated clinical study. A prospective, single arm unblinded, open label study will be carried out to determine the feasibility of recruitment, retention and adherence of 36 prostate cancer survivors who have been on androgen deprivation therapy within the last 5 years for a lifestyle modification intervention.

DETAILED DESCRIPTION:
INTRODUCTION:

Androgen deprivation therapy (ADT) has been demonstrated to improve disease free and over-all survival in men with prostate cancer (PCa).

ADT for PCa is associated with adverse cardio-metabolic effects such as reduced libido, hot flashes, metabolic syndrome, diabetes, myocardial infarction and stroke. This reduces quality of life (QoL) and potentially affects mortality.

There is paucity of data regarding comprehensive lifestyle interventions in men on ADT for Pca. Existing studies used non-standardized interventions or lack data on metabolic risk factors.

CLIPP is designed to address these gaps by using an intervention modelled after the Diabetes Prevention Program (DPP) with an emphasis on low carbohydrate and a Keto Diet, a standardized multi-component intervention with demonstrated effectiveness in reducing diabetes risk factors that has been successfully adapted for multiple disease types including breast cancer.

INTERVENTION:

* 24 Weeks
* Health Coaching Weekly
* Serum & Urine Baseline, Week 12 and Week 24
* Anthropometric Measures
* Questionnaires
* BMI Measurements

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer Stage I, II or III
* On androgen deprivation therapy with last 5 years
* Willing to participate in a lifestyle modification program
* Willing to modify diet and eating practices
* Willing to participate in blood collection, urine collection and measurements
* Minimum of 30 days since participating in another study/trial
* English speaking
* 40 to 80 years of age
* BMI >25%

Exclusion Criteria:

* Currently participating in another study or trial
* Currently in hospice
* Inability to walk two city blocks
* Inability to comprehend informed consent or procedural requirements
* Digestive Diseases (IBD, Diverticulitis, etc) that might prevent him from increasing fruit and vegetable intake
* Subjects already following an intensive lifestyle modification plan
* BMI <25%

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Reach Recruiting Target | 6 Months
  Recruit 36 men with prostate cancer who have been on androgen deprivation therapy within the last 5 years.
Retention of Participants | 6 Months
  75% retention rate
Adherence to Intervention | 6 Months
  75% attendance rate throughout 24 intervention visits

SECONDARY OUTCOMES:
Fasting Glucose | 6 Months
  Unit of Measure Mg/dL
Lipid Panel | 6 Months
  Unit of Measure Mg/dl
Hemoglobin A1c | 6 Months
  Unit of Measure %
CBC | 6 Months
  Unit of Measure Mg/dL
CMP | 6 Months
  Unit of Measure Mg/dL
Global Quality of Life Questionnaire | 6 Months
  PROMIS Scale v 1.2 Global Health. Scale Measurements 1 to 5 1=Poor 5=Excellent
Specific Quality of Life Questionnaire | 6 Months
  Expanded Prostate Cancer Index Composite Short Form (EPIC-26) Scale of Measurement 0 to 4. 0=No Problem 4=Big Problem

OTHER OUTCOMES:
Inflammatory Pathways Associated with Prostate Cancer | 6 Months
  Inflammation markers measured will include Interleukin-6, Interleukin 1-beta, Interleukin-8, stromal cell derived factor 1-alpha & basic fibroblast growth factor.
Angiogenic Pathways Associated with Prostate Cancer | 6 Months
  Determine the effect of comprehensive lifestyle modification intervention on angiogenesis, markers, important mechanisms for prostate cancer progression using blood, serum and urine. Angiogenesis markers will include vascular endothelial growth factor & plasma placental growth factor using Enzyme Linked Immunosorbent Assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Algotar, MD, PhD, MPH, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Algotar AM, Kumar R, Babiker HM, Dougherty ST, Hsu CH, Chow HH, Smith TE, Marrero DG, Courneya KS, Abraham I, Ligibel JA, Thomson CA. Protocol for a feasibility and early efficacy study of the Comprehensive Lifestyle Improvement Program for Prostate Cancer-2 (CLIPP2). Contemp Clin Trials Commun. 2021 Jan 13;21:100701. doi: 10.1016/j.conctc.2021.100701. eCollection 2021 Mar. PMID 33511299